CLINICAL TRIAL: NCT00870038
Title: Early Re-Endothelialization Might Not be the Unique Solution to Prevent Restenosis. The EREMUS Study
Brief Title: To Achieve an Early Reendothelialization at the Expense of Low Restenosis: The EREMUS Study
Acronym: EREMUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale della Misericordia (Other)
Responsible Party: Bernardo Cortese, Ospedale della Misericordia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bernard1
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-03

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Percutaneous Coronary Intervention
Keywords: PCI; stent; drug eluting stent; reendothelialization; restenosis; Percutaneous Coronary Angioplasty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Paclitaxel eluting balloon (Elutax) + Genous stent
  Interventions: Device: Percutaneous coronary intervention: Paclitaxel eluting balloon (Elutax) + Genous stent
- 2 (Experimental): Uncoated balloon + Genous stent
  Interventions: Device: Percutaneous coronary intervention: Uncoated balloon + Genous stent
- 3 (Active Comparator): Drug eluting stent (Taxus stent)
  Interventions: Device: Percutaneous coronary intervention: Drug eluting stent (Taxus stent)

INTERVENTIONS:
Device: Percutaneous coronary intervention: Paclitaxel eluting balloon (Elutax) + Genous stent — Predilatation with paclitaxel-eluting balloon, then stenting of the lesion with Genous stent
  Other Names: Elutax balloon, Aachen Resonance GmbH, Bavaria, Germany;; Genous stent, Orbus Neich, Fort Lauderdale, FL.
  Arms: 1
Device: Percutaneous coronary intervention: Uncoated balloon + Genous stent — Predilatation with uncoated balloon, the stenting with Genous stent.
  Other Names: Genous stent, Orbus Neich, Fort Lauderdale, FL.
  Arms: 2
Device: Percutaneous coronary intervention: Drug eluting stent (Taxus stent) — Predilatation with uncoated balloon, the placement of a Taxus stent.
  Other Names: Taxus stent, Boston Scientific, Natick, MA.
  Arms: 3

SUMMARY:
The investigators sought to discover which one of the following strategies is the safest for patients undergoing percutaneous coronary intervention: paclitaxel-coated balloon+Genous stent; Genous stent; drug eluting stent (paclitaxel).

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable angina pectoris suitable to PCI of at least one coronary vessel
* Age >18 years

Exclusion Criteria:

* Recent (<72 hours) acute myocardial infarction
* Creatinine clearance <40 ml/min
* Allergy or hypersensitivity to at least two between: aspirin, clopidogrel, heparin, bivalirudin, paclitaxel, contrast media
* Life expectancy <1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-08 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Late luminal loss between the three groups at 6 months angiographic follow up. | 6 months
Percent of stent struts covered by endothelium at optical coherence tomography, during 6 months angiographic follow up. | 6 months

SECONDARY OUTCOMES:
Angiographic restenosis (6 months angiographic follow up). | 6 months
Net adverse clinical events at 6 months (death, myocardial infarction, target lesion revascularization, bleedings as from Acuity scale). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Cortese, MD, FESC, Principal Investigator — Ospedale Maggiore Policlinico, Milano, Italy
Locations (1):
- U.O. Emodinamica, Ospedale della Misericordia, Grosseto, Italy

REFERENCES:
- [Result] Alfonso F, Zueco J, Cequier A, Mantilla R, Bethencourt A, Lopez-Minguez JR, Angel J, Auge JM, Gomez-Recio M, Moris C, Seabra-Gomes R, Perez-Vizcayno MJ, Macaya C; Restenosis Intra-stent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. A randomized comparison of repeat stenting with balloon angioplasty in patients with in-stent restenosis. J Am Coll Cardiol. 2003 Sep 3;42(5):796-805. doi: 10.1016/s0735-1097(03)00852-0. PMID 12957423
- [Result] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Result] Aoki J, Serruys PW, van Beusekom H, Ong AT, McFadden EP, Sianos G, van der Giessen WJ, Regar E, de Feyter PJ, Davis HR, Rowland S, Kutryk MJ. Endothelial progenitor cell capture by stents coated with antibody against CD34: the HEALING-FIM (Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth-First In Man) Registry. J Am Coll Cardiol. 2005 May 17;45(10):1574-9. doi: 10.1016/j.jacc.2005.01.048. PMID 15893169
- [Result] Co M, Tay E, Lee CH, Poh KK, Low A, Lim J, Lim IH, Lim YT, Tan HC. Use of endothelial progenitor cell capture stent (Genous Bio-Engineered R Stent) during primary percutaneous coronary intervention in acute myocardial infarction: intermediate- to long-term clinical follow-up. Am Heart J. 2008 Jan;155(1):128-32. doi: 10.1016/j.ahj.2007.08.031. Epub 2007 Nov 26. PMID 18082503
- [Result] Stone GW, White HD, Ohman EM, Bertrand ME, Lincoff AM, McLaurin BT, Cox DA, Pocock SJ, Ware JH, Feit F, Colombo A, Manoukian SV, Lansky AJ, Mehran R, Moses JW; Acute Catheterization and Urgent Intervention Triage strategy (ACUITY) trial investigators. Bivalirudin in patients with acute coronary syndromes undergoing percutaneous coronary intervention: a subgroup analysis from the Acute Catheterization and Urgent Intervention Triage strategy (ACUITY) trial. Lancet. 2007 Mar 17;369(9565):907-19. doi: 10.1016/S0140-6736(07)60450-4. PMID 17368152
- [Derived] Cortese B, Danzi GB, Piti A, Severi S, Limbruno U. Rationale and design of the randomized, multicenter EREMUS trial, a study that investigates how to achieve low restenosis and early reendothelialization after percutaneous coronary interventions. Catheter Cardiovasc Interv. 2011 Jul 1;78(1):32-7. doi: 10.1002/ccd.22856. Epub 2011 Mar 16. PMID 21413116